CLINICAL TRIAL: NCT00965484
Title: Multicenter, Open-Label Study Assessing Dyad (Subject And Caregiver) Perception Of Convenience And Preference Of The Newly Developed Mark VII Injection Pen
Brief Title: Genotropin Study Assessing Use of Injection Pen
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6281291
Record Dates: First submitted 2009-08-21; First posted 2009-08-25 (Estimated); Results first posted 2010-12-23 (Estimated); Last update posted 2011-01-28 (Estimated); Status verified 2010-04

CONDITIONS: Growth Hormone Deficiency; Idiopathic Short Stature
Keywords: Genotropin Medical device Patient reported outcome
MeSH Terms: conditions — Dwarfism, Pituitary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Genotropin pen (Experimental): All subjects will receive genotropin pen to use for 2 months.
  Interventions: Device: New Genotropin Pen

INTERVENTIONS:
Device: New Genotropin Pen — Subjects will use the genotropin pen for 2 months. After 2 months patients and caregiver will be asked to fill out a questionnaire to assess perception of the genotropin pen

SUMMARY:
Assessment of Genotropin patient and caregiver (Dyad) perception of convenience and preference of Genotropin injection pen. Patients already on genotropin will be asked to use a genotropin pen for 2 months. Patient and caregiver will be asked to complete a questionnaire at baseline and 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 8-18 years
* Using genotropin pen for at least 3 months prior to study enrollment
* Compliance with genotropin treatment

Exclusion Criteria:

* Medical conditions that can affect participation in study
* Insufficient command of English language to understand questionnaire
* Using other growth hormone device and not Genotropin pen

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 136 (Actual)
Dates: Start 2009-10; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (21):
- United States (21):
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Greenwood Village, Colorado
  - Pfizer Investigational Site, Gainesville, Florida
  - Pfizer Investigational Site, Tallahassee, Florida
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Southaven, Mississippi
  - Pfizer Investigational Site, Kansas City, Missouri
  - Pfizer Investigational Site, Morristown, New Jersey
  - Pfizer Investigational Site, Akron, Ohio
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Florence, South Carolina
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Fort Worth, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Seattle, Washington

REFERENCES:
- [Derived] Hey-Hadavi J, Pleil A, Deeb LC, Fuqua JS, Silverman LA, Reiner B, Newfield R, Rajicic N, Wajnrajch MP, Cara JF. Ease of use and preference for a new disposable self-injection pen compared with a reusable pen for administering recombinant human growth hormone: A multicenter, 2-month, single-arm, open-label clinical trial in patient-caregiver dyads. Clin Ther. 2010 Nov;32(12):2036-47. doi: 10.1016/j.clinthera.2010.11.007. PMID 21118739
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6281291&StudyName=Genotropin%20Study%20Assessing%20Use%20of%20Injection%20Pen

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who used the Genotropin® Pen for at least 3 months prior to enrollment were eligible to participate. Genotropin (somatropin) dose was not adjusted for the purposes of the study, but only based on clinical management requirements as determined by the treating physician.
Groups:
- Genotropin / Genotropin Mark VII Pen: Genotropin (somatropin) injection administered using the Genotropin Mark VII Pen subcutaneously (sc) at a dose prescribed by the physician.
Period: Overall Study
Arm/Group | Genotropin / Genotropin Mark VII Pen
Started | 136
Completed | 134
Not Completed | 2
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Genotropin / Genotropin Mark VII Pen
Number analyzed (Participants) | 136
Age, Customized [Number; unit: participants]
  ≤10 years of age | 37
  Between 11 and 12 years of age | 30
  Between 13 and 14 years of age | 40
  ≥15 years of age | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 91

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Dyads (Participant and Caregiver or Parent) Reporting no Difference or Easier to Use for New Genotropin Mark VII Injection Pen Compared to Pre-study Experience With the Genotropin Pen®
Description: Ease of use measured using the Injection Pen Assessment Questionnaire (IPAQ) patient-reported outcome (PRO) tool (based on 13 unique characteristics of injection pens). Section I measures ease of use of Genotropin® (very easy, somewhat easy, neither easy nor difficult, somewhat difficult, or very difficult). Section II measures ease of use of new Genotropin Mark VII Pen in comparison to pre-study experience with Genotropin® Pen (Genotropin® pen easier to use, new injection pen easier to use, or no difference) and preference (prefer Genotropin® Pen, prefer new injection pen, or no preference).
Time Frame: 2 months
Population: Full analysis set (FAS): all participants who used the new pen at least once to administer Genotropin and who completed the 2-month follow-up questionnaire. Dyad defined as the participant (child being treated) and adult partner (parent or caregiver).
Measure: Number (95% Confidence Interval); unit: percentage of dyads
Arm/Group | Genotropin / Genotropin Mark VII Pen
Number analyzed (Participants) | 133
percentage of dyads | 73.68 [66.20 to 81.17]

2. Secondary Outcome: Percentage of Dyads Reporting no Preference or Preference for New Genotropin Mark VII Injection Pen Compared to Pre-study Experience With the Genotropin Pen®
Description: Preference for use measured using IPAQ PRO tool (ease of use and preference based on 13 unique characteristics of injection pens). Section I measures ease of use of Genotropin® (very easy, somewhat easy, neither easy nor difficult, somewhat difficult, or very difficult). Section II measures ease of use of new Genotropin Mark VII Pen in comparison to pre-study experience with Genotropin® Pen (Genotropin® Pen easier to use, new injection pen easier to use, or no difference) and preference (prefer Genotropin® Pen, prefer new injection pen, or no preference).
Time Frame: 2 months
Population: FAS; N=number of participants with measurement.
Measure: Number (95% Confidence Interval); unit: percentage of dyads
Arm/Group | Genotropin / Genotropin Mark VII Pen
Number analyzed (Participants) | 132
percentage of dyads | 65.15 [57.02 to 73.28]

3. Secondary Outcome: Percentage of Dyads Reporting New Genotropin Mark VII Injection Pen Easier to Use Compared to Pre-study Experience With the Genotropin Pen®
Description: Ease of use measured using the IPAQ PRO tool (ease of use and preference based on 13 unique characteristics of injection pens). Section I measures ease of use of Genotropin® Pen (very easy, somewhat easy, neither easy nor difficult, somewhat difficult, or very difficult). Section II measures ease of use of new Genotropin Mark VII Pen in comparison to pre-study experience with Genotropin® Pen (Genotropin® Pen easier to use, new injection pen easier to use, or no difference) and preference (prefer Genotropin® Pen, prefer new injection pen, or no preference).
Time Frame: 2 months
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of dyads
Arm/Group | Genotropin / Genotropin Mark VII Pen
Number analyzed (Participants) | 133
percentage of dyads | 63.16 [54.96 to 71.36]

4. Secondary Outcome: Percentage of Dyads Reporting New Genotropin Mark VII Injection Pen Preferable Compared to Pre-study Experience With the Genotropin Pen®
Description: as for outcome 2
Time Frame: 2 months
Population: FAS; number of participants with measurement.
Measure: Number (95% Confidence Interval); unit: percentage of dyads
Arm/Group | Genotropin / Genotropin Mark VII Pen
Number analyzed (Participants) | 132
percentage of dyads | 59.85 [51.49 to 68.21]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Genotropin / Genotropin Mark VII Pen
Serious Adverse Events (participants affected / at risk) | 0/136
Other Adverse Events (participants affected / at risk) | 28/136
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Genotropin / Genotropin Mark VII Pen (N=136)
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Chills (General disorders) | 1
Influenza like illness (General disorders) | 1
Injection-site hematoma (General disorders) | 3 — Device related n=3
Injection-site pain (General disorders) | 5 — Device related n=5
Pyrexia (General disorders) | 4
Gastroenteritis viral (Infections and infestations) | 2
Gastrointestinal viral infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Pharyngitis streptococcal (Infections and infestations) | 3
Sinusitis (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 4
Animal scratch (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Joint sprain (Injury, poisoning and procedural complications) | 1
Limb injury (Injury, poisoning and procedural complications) | 1
Skin laceration (Injury, poisoning and procedural complications) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 7
Migraine (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.